CLINICAL TRIAL: NCT04843189
Title: Prospective Registration Study of Robtic Laparoscopy Versus Laparoscopy Assisted Colon Cancer Surgery
Acronym: STARS-CC02
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: The First Hospital of Jilin University (Other)
Responsible Party: Principal Investigator, Quan Wang, Professor, The First Hospital of Jilin University
Other Study IDs: STARS-CC02
Record Dates: First submitted 2021-04-06; First posted 2021-04-13 (Actual); Last update posted 2021-04-13 (Actual); Status verified 2021-04

CONDITIONS: Da Vinci Robot; Colon Cancer; Surgery
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Da Vinci Robotic Surgery Group: Da Vinci Robotic Surgery Group
  Interventions: Procedure: Da Vinci Robotic Surgery
- Laparoscopy-assisted surgery group: Laparoscopy-assisted surgery group
  Interventions: Procedure: Da Vinci Robotic Surgery

INTERVENTIONS:
Procedure: Da Vinci Robotic Surgery — Da Vinci Robotic Surgery

SUMMARY:
The purpose of this study is to compare the clinical data of patients with colon cancer who received robotic or laparoscopic surgery, and to compare the short-term and long-term effects of robotic surgery in the treatment of colon cancer. To verify the safety and effectiveness of the corresponding surgical methods, and provide better guidance for the following clinical practice.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18-80 years old, male or female;
2. Colon cancer (ascending colon, transverse colon, descending colon, sigmoid colon) is diagnosed by histology or cytology;
3. The clinical stage is T1-4aN0-2M0; 4 No multiple distant metastases;

5. ECOG score 0-2; 6. Heart, lung, liver, and kidney functions can tolerate surgery; 7. Patients and their families can understand and are willing to participate in this clinical study, and sign an informed consent.

Exclusion Criteria:

1. Past history of malignant colorectal tumors or recent diagnosis combined with other malignant tumors;
2. Patients with intestinal obstruction, intestinal perforation, intestinal bleeding, etc. who need emergency surgery;
3. Neighboring organs need to be combined with organ resection;
4. New adjuvant therapy before surgery;
5. ASA grade ≥ grade IV and/or ECOG physical status score> 2 points;
6. Those who have severe liver and kidney function, cardiopulmonary function, blood coagulation dysfunction, or combined with serious underlying diseases that cannot tolerate surgery;
7. Have a history of severe mental illness;
8. Pregnant or lactating women;
9. Patients with other clinical and laboratory conditions considered by the investigator should not participate in the trial.

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with colon cancer
Sampling Method: Probability Sample
Enrollment: 648 (Estimated)
Dates: Start 2021-05-01 (Estimated); Primary Completion 2023-05-01 (Estimated); Study Completion 2023-05-01 (Estimated)

PRIMARY OUTCOMES:
Number of lymph nodes harvested | During the operation
  Number of lymph nodes harvested

SECONDARY OUTCOMES:
Operation time | During the operation
  Operation time
Length of surgical incision | During the operation
  Length of surgical incision
Intraoperative blood loss | During the operation
  Intraoperative blood loss
Intraoperative concversion rate | During the operation
  Intraoperative concversion rate
Postoperative recovery | During the postoperative hospital stay
  first exhaust, defecation time, restoring liquid diet, hospitalization days, etc.
3-year disease-free survival | 3 years after surgery
  3-year disease-free survival
5-year overall survival | 5 years after surgery
  5-year overall survival

CONTACTS AND LOCATIONS:
Locations (1):
- Jilin University First Hospital, Changchun, Jilin, China

IPD SHARING:
Plan to Share IPD: No